CLINICAL TRIAL: NCT01588795
Title: Renal Denervation in Patients With Diabetic Nephropathy and Persistent Proteinuria
Brief Title: Renal Denervation in Diabetic Nephropathy
Acronym: DERENEDIAB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P110122
Record Dates: First submitted 2012-04-18; First posted 2012-05-01 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Diabetic Nephropathy; Persistent Proteinuria With Type II Diabetes
Keywords: Diabetic nephropathy; renal denervation; nephroprotection; Renal failure; Renal injury; End stage renal disease
MeSH Terms: conditions — Diabetic Nephropathies; Renal Insufficiency; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Denervation + TMNS (Experimental): Patients are treated with the renal denervation procedure after randomization and are maintained on standardized anti-proteinuric medications
  Interventions: Procedure: Percutaneous renal denervation and TMNS
- TMNS (Active Comparator): Patients are maintained on standardized anti-proteinuric medications
  Interventions: Drug: Standardized antiproteinuric medication regimen includes an angiotensin receptor blocker , a diuretic , 25OH vitamin D3 and a statin

INTERVENTIONS:
Procedure: Percutaneous renal denervation and TMNS — Patients are treated with the renal denervation procedure after randomization and are maintained on standardized anti-proteinuric medications
  Arms: Denervation + TMNS
Drug: Standardized antiproteinuric medication regimen includes an angiotensin receptor blocker , a diuretic , 25OH vitamin D3 and a statin — Patients are maintained on Standardized antiproteinuric medication regimen includes an angiotensin receptor blocker (irbesartan 300mg), a diuretic (furosemide 40mg or indapamide LP 1.5mg according to the eGFR), 25OH vitamin D3 and a statin (atorvastatin 20mg)
  Arms: TMNS

SUMMARY:
The DERENEDIAB study is a proof-of-concept, multi-center, prospective, open, randomized, controlled study of the effectiveness of renal denervation in addition to standardized medical treatment compared to medical treatment alone in diabetic subjects with diabetic nephropathy and resistant proteinuria. Bilateral renal denervation will be performed using the Symplicity Catheter - a percutaneous system that delivers radiofrequency (RF) energy through the luminal surface of the renal artery.

DETAILED DESCRIPTION:
The DERENEDIAB study is a proof-of-concept multi-center, prospective, open, randomized, controlled study of the effectiveness of renal denervation in addition to standardized medical treatment compared to medical treatment alone in diabetic subjects with diabetic nephropathy and resistant proteinuria. Bilateral renal denervation will be performed using the Symplicity Catheter - a percutaneous system that delivers radiofrequency (RF) energy through the luminal surface of the renal artery.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus male or female patient
* Individual is > 18 and ≤ 75 years old
* Diabetic nephropathy (if no pathological examination, diagnosis based on the association of history of diabetes, diabetic retinopathy and no hematuria)
* Proteinuria/creatininuria ratio > 0.1 g/mmol lasting for 8 weeks
* Under stable medication regimen including for at least 2 months full tolerated doses of al least 1 RAAS blocker (ACEI, renin inhibitor, ARB) and a diuretic
* 2 functional kidneys sizing ≥ 90 mm; eGFR > 20 mL/min/1.73m² (MDRD formula
* Suitable aorto-renal vascular anatomy compatible with the endovascular denervation procedure; Informed consent has been signed
* Health insurance policy active

Exclusion Criteria:

* Patients with an estimated glomerular filtration rate (eGFR) of less than 20 mL/min/1.73 m2
* Patients unable to sign an informed consent, to understand the protocol, living too far from the specialized center
* Non-diabetic renal disease
* Patients with severe hypertension (grade 3 ESH classification)
* Kaliemia ≥ 6mmol/L
* History of nephrogenic fibrosis-induced MRI contrast media
* Patient with single functioning kidney
* Patient with contrast media allergy
* Patient with any implantable device incompatible with low frequency waves delivery
* Patient with contra-indication to the anti-proteinuric standardized medication regimen
* Patient with transient or fixed cerebral ischemia within 3 months before inclusion
* Patient with myocardial infarction, unstable angina pectoris, coronary bypass or percutaneous angioplasty within 3 months before inclusion
* Patient with asthma or chronic obstructive pulmonary disease with a contra-indication to beta-blockers medication
* Patient with type 1 diabetes mellitus
* Uncontrolled type 2 diabetes mellitus (Hb1Ac > 10%)
* Patient with malignancy within the 5 past years
* Patient with any medical or surgical condition that could worsen the risk of the study, according to the investigator; Patient with chronic alcohol consumption
* Patient with atrial fibrillation and/or a brachial circumference of ≥ 42cm
* Patient is pregnant, nursing or planning to be pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
proteinuria/creatininuria ratio | from baseline to 1 year

SECONDARY OUTCOMES:
Number of patients with a decrease of the PU/CrU >50% ratio | from baseline to 1 year
Evaluation of the slope of decay of the PU/CrU | from baseline to 1 year
eGFR is estimated by the MDRD formula, and is expressed in mL/min/1.73m². The direct GFR will be assessed by measuring the 51Cr-EDTA plasmatic clearance | from baseline to 1 year
  eGFR is estimated by the MDRD formula, and is expressed in mL/min/1.73m². The direct GFR will be assessed by measuring the 51Cr-EDTA plasmatic clearance
Outcome of the GFR assessed by 51Cr-EDTA clearance | from randomisation to 1 year
  Only in the experimental arm
Decrease of the blood pressure assessed on ABPM | From randomisation to 1 year
Anti-hypertensive regimen score | from baseline to 1 year
Evaluation of the renal arterial anatomy | from baseline to 1 year
  in the experimental group:number of principal renal artery. Should be 1/ kidney of at least 4mm diameter and 10mm long. One accessory artery is acceptable if <
Evaluation of safety and tolerance of renal denervation in diabetic patients with overt proteinuria | from baseline to 1 year
  in the experimental group:Occurrence of adverse events: acute renal failure, damage on the renal artery (dissection, perforation, thrombosis), allergy to the contrast media, worsening of any dysautonomia
Evaluate the outcome of biological parameters | from baseline to 1 year
  eGFR (MDRD formula), proteinuria/creatininuria ratio
Evaluate the diabetic neuropathy/dysautonomy | from randomisation to 1 year
  in the experimental:blood pressure in orthostatism, pulse wave velocimetry, RR interval on the Holter ECG, cutaneous baroreflex
Evaluate the outcome of specific kidney injury markers | from randomisation to 1 year
  in the experimental group:urinary levels of KIM1 and NGAL before and 1 year after the denervation

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Bobrie, MD, Principal Investigator — HTA department
Locations (1):
- CIC Hopital europeen george pompidou, Paris, Paris, France

REFERENCES:
- [Derived] Persu A, Sapoval M, Azizi M, Monge M, Danse E, Hammer F, Renkin J. Renal artery stenosis following renal denervation: a matter of concern. J Hypertens. 2014 Oct;32(10):2101-5. doi: 10.1097/HJH.0000000000000323. No abstract available. PMID 25186534